CLINICAL TRIAL: NCT02582151
Title: A Randomized Trial of Transcutaneous Nerve Stimulation for Neurogenic Bladder
Brief Title: Transcutaneous Peripheral Neuromodulation for Neurogenic Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 107210
Record Dates: First submitted 2015-10-13; First posted 2015-10-21 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Urinary Bladder, Neurogenic
MeSH Terms: conditions — Urinary Bladder, Neurogenic | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham tibial nerve stimulation (Sham Comparator): Use of peripheral nerve stimulator in a location that will not actively stimulate the tibial nerve.
  Interventions: Device: EV-906 Digital Transcutaneous electrical nerve stimulation (TENS) machine
- Tibial nerve stimulation (Active Comparator): Transcutaneous peripheral nerve stimulator in a location that will actively stimulate the tibial nerve.
  Interventions: Device: EV-906 Digital Transcutaneous electrical nerve stimulation (TENS) machine

INTERVENTIONS:
Device: EV-906 Digital Transcutaneous electrical nerve stimulation (TENS) machine — Percutaneous patch electrodes are used to deliver low level electrical currents.

SUMMARY:
Neurogenic bladder patients may have symptoms of urinary frequency, urgency, urgency incontinence and voiding symptoms due to bladder dysfunction arising from their underlying neurologic condition. Current treatment options are effective for some patients, however many patients are not optimally managed due to modest efficacy or significant side effects. Second line therapies include intravesical onabotulinum toxin, however it is associated with a risk of urinary retention, and patients with neurologic disorders often are unable to perform self catheterize due to physical limitations. Sacral neuromodulation is associated with an undesirably high cost and potential complications in this population. The use of transcutaneous tibial nerve stimulation is an alternative form of neuromodulation, and it may have some potential benefits over percutaneous tibial nerve stimulation. While some preliminary studies have suggested it may be effective, there are no high quality randomized trials. This proposal is a 3 month, randomized, sham-controlled, clinical trial to evaluate the short term clinical efficacy of at home transcutaneous tibial nerve stimulation. Valid and reliable patient reported outcome measures, and objective measures of incontinence have been included as outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age, with a clinical condition associated with neurogenic bladder dysfunction (multiple sclerosis, Parkinson's disease, stroke, dementia, cerebral palsy, spinal cord injury)(27).
2. Failure of behavioral measures and/or pharmacologic therapy to adequately control neurogenic bladder symptoms.

Exclusion Criteria:

1. Current or previous percutaneous/transcutaneous tibial nerve stimulation or sacral neuromodulation therapy
2. Stress predominant urinary incontinence
3. Newly added bladder medication or dose change with the last 2 months (Tamsulosin, Silodosin, Alfuzosin, Terazosin, Baclofen, Diazepam, amitriptyline, imipramine, DDAVP, tolterodine, oxybutynin, fesoterodine, darifenacin, solifenacin, trospium, mirabegron)
4. Intravesical botulinum toxin use within the last 1 year
5. Implanted pacemaker or defibrillator
6. History of epilepsy
7. Unable or unwilling to commit to study treatment schedule
8. Pregnant, or possible pregnancy planned for the duration of the study period
9. Active skin disease of the lower legs (dermatitis, cellulitis, eczema, trauma)
10. Documented allergy to patch electrodes or their adhesive
11. Metallic implant within the lower limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham Tibial Nerve Stimulation | Tibial Nerve Stimulation
Started | 14 | 16
Completed | 12 | 16
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Tibial Nerve Stimulation | Tibial Nerve Stimulation | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [44 to 60] | 60 [49 to 65] | 56 [47 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Patient Perception of Bladder Condition Questionnaire
Description: Patient perception of bladder condition (PPBC) question. It is scored from 0 (My bladder condition does not cause me any problems at all) to 5 (My bladder condition causes me many severe problems). Higher numbers are worse outcomes.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Sham Tibial Nerve Stimulation | Tibial Nerve Stimulation
Number analyzed (Participants) | 14 | 16
units on a scale | 3 [3 to 3] | 3 [2 to 4]

2. Secondary Outcome: Neurogenic Bladder Symptom Score (NBSS) Questionnaire
Description: The NBSS is a patient reported symptom score covering three domains: incontinence, storage/voiding, and consequences. It is scored from 0 to 72, and a higher score is worse outcome.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Sham Tibial Nerve Stimulation | Tibial Nerve Stimulation
Number analyzed (Participants) | 14 | 16
Units on a scale | 33 [29 to 38] | 29 [25 to 33]

3. Secondary Outcome: Qualiveen-Short Form Questionnaire
Description: Patient reported questionnaire that measures quality of life among neurogenic bladder patients. Score ranges from 0 to 32. A higher score is worse.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Sham Tibial Nerve Stimulation | Tibial Nerve Stimulation
Number analyzed (Participants) | 14 | 16
units on a scale | 27 [23 to 31] | 27 [24 to 31]

4. Secondary Outcome: 3-day Voiding Diary
Description: Daily urinary frequency as recorded by the patient over 3 days. Summarised as an average daily frequency.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: voids per 24 hrs
Arm/Group | Sham Tibial Nerve Stimulation | Tibial Nerve Stimulation
Number analyzed (Participants) | 14 | 16
voids per 24 hrs | 9 [8 to 11] | 9 [7 to 10]

5. Secondary Outcome: 24hr Incontinence Pad Weights
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | Sham Tibial Nerve Stimulation | Tibial Nerve Stimulation
Number analyzed (Participants) | 14 | 16
grams | 364 [333 to 395] | 362 [334 to 391]

6. Secondary Outcome: Physician Assessment of Patient Benefit (Global Response Scale)
Description: Completed by physicians based on their assessment after discussion with the patient as to the amount of benefit they received. Reported on a scale of 0 (no benefit) to 7 (substantial benefit)
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Sham Tibial Nerve Stimulation | Tibial Nerve Stimulation
Number analyzed (Participants) | 14 | 16
units on a scale | 3 [3 to 3] | 3 [2 to 3]

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Sham Tibial Nerve Stimulation | Tibial Nerve Stimulation
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT02582151/Prot_SAP_000.pdf